CLINICAL TRIAL: NCT07305350
Title: EFFICACY OF MELATONIN IN MANAGEMENT OF HYPOXIC ISCHEMIC ENCEPHALOPATHY (HIE) IN NEONATES
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Child Health Sciences and Children's Hospital, Lahore (Other)
Responsible Party: Principal Investigator, Dr. Amina Cheema, Dr Amina Cheema, University of Child Health Sciences and Children's Hospital, Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No/779/CH-UCHS
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Hypoxic Ischaemic Encephalopathy (HIE)
Keywords: Hypoxic ischemic encephalopathy (HIE); Melatonin; Randomized Control Trial
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Melatonin; Fluid Therapy

STUDY DESIGN:
Intervention Model Description: It is a Randomized control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): 55 neonates will be assigned group A in which newborns will be given single 10mg dose of melatonin through nasogastric tube in addition to standard supportive therapy.
  Interventions: Drug: Melatonin
- Group B (Active Comparator): 55 neonates will be assigned group B in which patients will be given standard supportive therapy only. Standard supportive therapy included oxygen therapy, intravenous (IV) fluids, intensive monitoring, broad-spectrum antibiotic cover for possible role of infection
  Interventions: Combination Product: intravenous (IV) fluids, intensive monitoring, broad-spectrum antibiotic cover

INTERVENTIONS:
Drug: Melatonin — 55 neonates will be assigned group A in which newborns will be given single 10mg dose of melatonin through nasogastric tube in addition to standard supportive therapy.
  Arms: Group A
Combination Product: intravenous (IV) fluids, intensive monitoring, broad-spectrum antibiotic cover — 55 neonates will be assigned group B in which patients will be given standard supportive therapy only.
  Arms: Group B

SUMMARY:
To compare the survival rate and improvement in stage of hypoxic ischemic encephalopathy (HIE) at day 7 of treatment in neonates treated with versus without melatonin in addition to standard supportive therapy.

DETAILED DESCRIPTION:
This is a randomized control trial and the purpose of this study is to determine efficacy of melatonin in management of hypoxic ischemic encephalopathy in newborns. Baseline characteristics will be documented after which patients will be divided into two groups by paper lottery method namely group A in which newborns will be given single 10mg dose of melatonin through nasogastric tube in addition to standard supportive therapy and group B in which patients will be given standard supportive therapy only.

ELIGIBILITY:
Inclusion criteria:

All term infants (as per operational definition). Both genders. Presenting with hypoxic ischemic encephalopathy (as per operational definition).

Exclusion criteria:

Drug reactions. Newborns at gestational age < 36 weeks. Neonates whose mother received general anesthesia. Neonates with congenital malformations. Neonates whose mother received anticonvulsants. Neonates not fulfilling criteria for HIE. Neonatal sepsis, pneumonia or in-born error of metabolism.

Min Age: 1 Hour | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-05-10 (Estimated); Study Completion 2026-05-10 (Estimated)

PRIMARY OUTCOMES:
Neonate survival rate | 28 days of life
  Role of melatonin will be determined primarily by survival rate in neonates with hypoxic ischemic encephalopathy at 28 days of life.

SECONDARY OUTCOMES:
Improvement in stage of HIE | Day 1, 3 and 7 of life
  Secondary outcome measures to determine role will be improvement in stage of hypoxic ischemic encephalopathy (based on Thomson score) at day 1, 3 and 7.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Khalid Masood, MBBS, FCPS, Study Chair — Children Hospital and University of Child Health Sciences, Lahore
Locations (1):
- Children Hospital and University of Child Health Sciences, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Due to confidentiality

REFERENCES:
- [Background] Siddiqui MA, Butt TK. Role of Intravenous Magnesium Sulphate in Term Neonates with Hypoxic Ischemic Encephalopathy (HIE) in a Low-income Country: A Randomised Clinical Trial. J Coll Physicians Surg Pak. 2021 Jul;31(7):817-820. doi: 10.29271/jcpsp.2021.07.817. PMID 34271782
- [Background] Ran Y, Ye L, Ding Z, Gao F, Yang S, Fang B, Liu Z, Xi J. Melatonin Protects Against Ischemic Brain Injury by Modulating PI3K/AKT Signaling Pathway via Suppression of PTEN Activity. ASN Neuro. 2021 Jan-Dec;13:17590914211022888. doi: 10.1177/17590914211022888. PMID 34120482
- [Background] Packer CH, Hersh AR, Sargent JA, Caughey AB. Therapeutic hypothermia in severe hypoxic-ischemic encephalopathy: a cost-effectiveness analysis. J Matern Fetal Neonatal Med. 2022 Mar;35(5):890-897. doi: 10.1080/14767058.2020.1733519. Epub 2020 Mar 10. PMID 32156180
- [Background] Michniewicz B, Al Saad SR, Karbowski LM, Gadzinowski J, Szymankiewicz M, Szpecht D. Organ Complications of Infants with Hypoxic Ischemic Encephalopathy Before Therapeutic Hypothermia. Ther Hypothermia Temp Manag. 2021 Mar;11(1):58-63. doi: 10.1089/ther.2020.0035. Epub 2020 Nov 5. PMID 33155883
- [Background] Iqbal N, Younus J, Malik M, Fatima B, Imran A, Maqbool S, Irfan Waheed KA, Haque K. The Neuroprotective Efficacy of Postnatal Magnesium Sulfate in Term or Near-Term Infants With Moderate-to-Severe Birth Asphyxia. Cureus. 2021 Aug 2;13(8):e16826. doi: 10.7759/cureus.16826. eCollection 2021 Aug. PMID 34513419
- [Background] Go H, Saito Y, Maeda H, Maeda R, Yaginuma K, Ogasawara K, Kashiwabara N, Kawasaki Y, Hosoya M. Serum cytokine profiling in neonates with hypoxic ischemic encephalopathy. J Neonatal Perinatal Med. 2021;14(2):177-182. doi: 10.3233/NPM-200431. PMID 33074195
- [Background] Florido J, Rodriguez-Santana C, Martinez-Ruiz L, Lopez-Rodriguez A, Acuna-Castroviejo D, Rusanova I, Escames G. Understanding the Mechanism of Action of Melatonin, Which Induces ROS Production in Cancer Cells. Antioxidants (Basel). 2022 Aug 20;11(8):1621. doi: 10.3390/antiox11081621. PMID 36009340
- [Background] Dolan F, Wintermark P. Updates in Treatment of Hypoxic-Ischemic Encephalopathy. Clin Perinatol. 2025 Jun;52(2):321-343. doi: 10.1016/j.clp.2025.02.010. Epub 2025 Mar 21. PMID 40350214
- [Background] Cornet MC, Kuzniewicz M, Scheffler A, Forquer H, Hamilton E, Newman TB, Wu YW. Perinatal Hypoxic-Ischemic Encephalopathy: Incidence Over Time Within a Modern US Birth Cohort. Pediatr Neurol. 2023 Dec;149:145-150. doi: 10.1016/j.pediatrneurol.2023.08.037. Epub 2023 Aug 31. PMID 37883841
- [Background] Chakkarapani E, de Vries LS, Ferriero DM, Gunn AJ. Neonatal encephalopathy and hypoxic-ischemic encephalopathy: the state of the art. Pediatr Res. 2025 Mar 24. doi: 10.1038/s41390-025-03986-2. Online ahead of print. PMID 40128590
- [Background] Bobba PS, Malhotra A, Sheth KN, Taylor SN, Ment LR, Payabvash S. Brain injury patterns in hypoxic ischemic encephalopathy of term neonates. J Neuroimaging. 2023 Jan;33(1):79-84. doi: 10.1111/jon.13052. Epub 2022 Sep 26. PMID 36164277
- [Background] Ahmad QM, Chishti AL, Waseem N. Role of melatonin in management of hypoxic ischaemic encephalopathy in newborns: A randomized control trial. J Pak Med Assoc. 2018 Aug;68(8):1233-1237. PMID 30108392
- [Background] Ahmed J, Pullattayil S AK, Robertson NJ, More K. Melatonin for neuroprotection in neonatal encephalopathy: A systematic review & meta-analysis of clinical trials. Eur J Paediatr Neurol. 2021 Mar;31:38-45. doi: 10.1016/j.ejpn.2021.02.003. Epub 2021 Feb 11. PMID 33601197